CLINICAL TRIAL: NCT03156322
Title: Effects of Different Epidural Initiation Volumes on Postoperative Analgesia in Cesarean Delivery
Brief Title: Different Epidural Initiation Volumes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Osman Kacmaz, Anesthesiologist, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Inonu Anesthesia
Record Dates: First submitted 2017-05-09; First posted 2017-05-17 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-05

CONDITIONS: Pain, Postoperative
Keywords: cesarean section; combined spinal epidural anesthesia; patient controlled epidural analgesia; postoperative pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine; Fentanyl

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 5 (Active Comparator): 5 mL epidural initiation volume (bupivacaine + fentanyl)
  Interventions: Drug: 5 mL epidural initiation volume (bupivacaine + fentanyl)
- Group 10 (Active Comparator): 10 mL epidural initiation volume (bupivacaine + fentanyl)
  Interventions: Drug: 10 mL epidural initiation volume (bupivacaine + fentanyl)
- Group 20 (Active Comparator): 20 mL epidural initiation volume (bupivacaine + fentanyl)
  Interventions: Drug: 20 mL epidural initiation volume (bupivacaine + fentanyl)

INTERVENTIONS:
Drug: 5 mL epidural initiation volume (bupivacaine + fentanyl) — 5 mL 0.625% bupivacaine + 2 μg/mL fentanyl solution is administered from epidural catheter
  Other Names: Bupivacaine(Marcaine 0.5%), Fentanyl(Talinat 0.5mg/10mL)
  Arms: Group 5
Drug: 10 mL epidural initiation volume (bupivacaine + fentanyl) — 10 mL 0.625% bupivacaine + 2 μg/mL fentanyl solution is administered from epidural catheter
  Other Names: Bupivacaine(Marcaine 0.5%), Fentanyl(Talinat 0.5mg/10mL)
  Arms: Group 10
Drug: 20 mL epidural initiation volume (bupivacaine + fentanyl) — 20 mL 0.625% bupivacaine + + 2 μg/mL fentanyl solution is administered from epidural catheter
  Other Names: Bupivacaine(Marcaine 0.5%), Fentanyl(Talinat 0.5mg/10mL)
  Arms: Group 20

SUMMARY:
The aim of this study is to compare the effect of different epidural initiation volumes on postoperative pain scores, local anesthetic requirements, and motor block in patients who undergo patient controlled epidural analgesia for postoperative pain after cesarean section.

DETAILED DESCRIPTION:
90 minutes after combined epidural spinal catheter insertion, three different volumes (5 mL, 10 mL, and 20 mL) are administered with a patient-controlled epidural analgesia (PCEA) device through the epidural catheter. For each group, 0.625% bupivacain + 2 μg/mL fentanyl, is administered.

The visual analog scale, first analgesic demand time, the number of PCEA requirement per hour, morphine requirement, nausea-vomiting, itching, motor block, hypotension, and total consumed analgesic, and ephedrine amounts of the patients are recorded in the recovery room and at postoperative 2, 4, 6, 12 hours.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology risks classification II
* Term pregnant

Exclusion Criteria:

* Multiple pregnancy
* Diabetes mellitus
* Hypertension
* Coagulopathy
* Severe cardiac, neurological and pulmonary disease
* Allergy to the study drugs
* Difficulty in understanding the use of the patient controlled analgesia device

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Change in postoperative pain scores | up to 12 hours after cesarean delivery
  Visual analog scale

SECONDARY OUTCOMES:
First analgesic demand time | up to 12 hours after cesarean delivery
  Time to first analgesic requirement (first patient controlled epidural analgesic demand time)
The number of analgesic requirement | up to 12 hours after cesarean delivery
  The number of patient controlled epidural analgesic requirement per hour
Morphine requirement | up to 12 hours after cesarean delivery
  Intravenous morphine administration

OTHER OUTCOMES:
Side effects associated with epidural analgesia | up to 12 hours after cesarean delivery
  Nausea-vomiting, itching, motor block, hypotension

CONTACTS AND LOCATIONS:
Overall Officials: Mahmut Durmus, Prof, Study Chair — Prof Dr
Locations (1):
- Inonu University Turgut Ozal Medical Center, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Sng BL, Woo D, Leong WL, Wang H, Assam PN, Sia AT. Comparison of computer-integrated patient-controlled epidural analgesia with no initial basal infusion versus moderate basal infusion for labor and delivery: A randomized controlled trial. J Anaesthesiol Clin Pharmacol. 2014 Oct;30(4):496-501. doi: 10.4103/0970-9185.142842. PMID 25425774